CLINICAL TRIAL: NCT06007820
Title: Efficacy & Safety of Pigtail Catheter Drainage Versus Need Based Thoracocentesis for Recurrent Hepatic Hydrothorax. A Randomized Controlled Trial
Brief Title: Efficacy & Safety of Pigtail Catheter Drainage Versus Need Based Thoracocentesis for Recurrent Hepatic Hydrothorax.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-60
Record Dates: First submitted 2023-08-05; First posted 2023-08-23 (Actual); Last update posted 2023-08-23 (Actual); Status verified 2023-08

CONDITIONS: Hepatic Hydrothorax

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Large Volume Thoracocentesis (Experimental): Group 1 - on-demand therapeutic thoracocentensis
  Interventions: Procedure: Large Volume Thoracocentesis
- Pigtail Catheter (Active Comparator): Group 2 - small volume frequent thoracocentesis using PCD
  Interventions: Procedure: Pigtail Catheter

INTERVENTIONS:
Procedure: Large Volume Thoracocentesis — Large Volume Thoracocentesis
  Arms: Large Volume Thoracocentesis
Procedure: Pigtail Catheter — Pigtail Catheter
  Arms: Pigtail Catheter

SUMMARY:
In cirrhotic patients with recurrent hepatic hydrothorax liver transplantation is a definitive treatment. But a significant number of individual are ineligible for liver transplantation. In these patients to ameliorate the symptoms various treatment modalities such as TIPS, serial thoracocentesis, pigtail catheter drainage and pleurodesis are used. We are doing this study to assess the safety and efficacy of serial thoracocentesis verus pigtail catheter drainage.

DETAILED DESCRIPTION:
* Study population - Cirrhotic patients with recurrent hepatic hydrothorax
* Study design - A prospective, randomized, single center open label study
* Block Randomization, block size - 10
* Sample size - Assuming in single time thoracocentesis group 5+/-3.67 thoracocentesis is required, investigator expect a 50 % reduction in pigtail drainage group. Apha error- 5, power -90, 15% dropout 35 patients in each arm
* Intervention - Group 1 - on-demand therapeutic thoracocentensis, Group 2 - small volume frequent thoracocentesis using PCD.
* Monitoring and assessment
* At enrollment:

(A) Complete history and examination

1. Etiology of cirrhosis
2. Severity of ascites, Jaundice
3. Prior Hepatic encephalopathy, bleed, Jaundice
4. Prior Spontaneous bacterial peritonitis, large volume paracentesis frequency
5. Pattern and number of prior decompensation
6. Prior Acute on Chronic Liver Failure and Acute Kidney episodes
7. Use of non selective beta blockers, norfloxaxin, rifaximin and albumin
8. History of Endoscopic Variceal ligation or other endotherapy
9. History of Hypertension, Diabetes
10. Fever , signs of sepsis (SIRS)
11. Examination- Sarcopenia, fraility, icterus, pedal edema

At follow-up (at daily till Day - 7, thereafter at Day - 30 and Day 90) Complete history and examination

1. Complications - SBP, SBE, ACLF and Jaundice, HE/ AKI episodes
2. HTN, Diabetes control
3. Fever , signs of sepsis (SIRS)
4. Examination- Sarcopenia, fraility, icterus, pedal edema, ascites, HE Clinical Evaluation

1. Etiology of chronic liver disease (Baseline) 2. Severity of liver disease (Baseline, Day - 7, Day - 30, Day - 90 ) 3. MELD score, MELD-Na score, CTP score (Baseline, Day - 7, Day - 30, Day - 90 ) 4. Complications (Baseline, Day - 7, Day - 30, Day - 90 ) 5. Overt HE, PHT related Bleed, clinical jaundice, ascites, hyponatremia, AKI, SBP, Infection (specify site and severity), Frequency of Large Volume Paracentesis, On Demand Thoracocentesis

* Labs and follow up Baseline (at admission) -

  1. Blood : KFT, LFT, CBC, INR, AFP, PCT, S.PRA, Pro-BNP, Urinary Na
  2. Imaging : USG abdomen, X-ray chest, 2D ECHO
  3. Pleural fluid/ ascitic fluid - TLC, DLC, Protein, Sugar, SPAG, SAAG, ADA, c/s
  4. Hemodynamics : Intrapleural pressures at first TT
  5. Baseline (at randomization, Day -3 and Day - 7 in PCD-TT) -
  6. Blood : KFT, INR; S.PRA, Pro-BNP, Urinary Na (at Day 7)
  7. Imaging : X-ray chest
  8. Pleural fluid/ ascitic fluid - TLC, DLC, SPAG, c/s if indicated
  9. Day - 60, Day - 90 (end of follow-up)
  10. Blood : KFT, LFT, CBC, INR, AFP
  11. Imaging : USG abdomen, X-ray chest, 2D ECHO
* STATISTICAL ANALYSIS -

  1. Data will be reported as mean + SD.
  2. Categorical variables will be compared using the chi-square test or Fisher exact test
  3. Normal continuous variables will be compared using the Student's t test
  4. Non normal continuous variables will be compared using the Mann-Whitney rank-sum test (unpaired data) or the Wilcoxon test (paired data).
  5. The actuarial probability of survival will be calculated by the Kaplan-Meier method and compared using the log-rank test.
  6. A Cox regression analysis will be performed to identify independent prognostic factors for survival.
  7. Univariate and multivariate analysis will be used whenever applicable.
* Adverse effects - Chest pain, pain at the site, Breathlessness, infection, pneumothorax, infection, bleeding
* Stopping rule -

  1. Liver Transplant
  2. Appearance of SBP, PICD, HE.
  3. Mortality
  4. End of follow-up

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years
2. CLD with refilling symptomatic hepatic hydrothorax

Exclusion Criteria:

1. CTP >12, MELD>25
2. Tubercular PE, Ischemic cardiac disease
3. If opting for TIPS/ LT
4. Severe HPS
5. Prior or current SBE/ SBP, septic shock
6. Patients on mechanical ventilator
7. Serum Creatinine >2 mg/dl
8. Extrahepatic malignancy
9. Serum Sodium < 120
10. Post TIPS/ BRTO/ SAE patients
11. Post renal or liver transplantation
12. Lack of informed consent
13. Hepatocellular carcinoma outside milan criteria
14. Non-cirrhotic portal HT
15. Known HIV infection
16. Pregnant women

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-08-15 (Estimated); Primary Completion 2024-02-27 (Estimated); Study Completion 2024-02-27 (Estimated)

PRIMARY OUTCOMES:
Frequency of Repeated Thoracocentesis | Day 30
Frequency of Repeated Thoracocentesis | Day 90

SECONDARY OUTCOMES:
Incidence of refilling hydrothorax within | 72 hours
Frequency of Repeated Thoracocentesis. | Day 30 and Day 90
Rate of Complete Response, Partial Response, No response. | Day 7, Day 30, Day 90
Number of times Thoracocentesis is required between both groups at Day 30 | Day 30
Number of times Thoracocentesis is required between both groups at Day 90 | Day 90
Proportion of pateint developing Post thoracocentesis Shock (Change in Heart Rate, Blood pressure) at Day 7 | Day 7
Proportion of pateint developing Post thoracocentesis Shock (Change in Heart Rate, Blood pressure) at Day 30 | Day 30
Proportion of pateint developing Post thoracocentesis Shock (Change in Heart Rate, Blood pressure) at Day 90 | Day 90
Change in Renal parameters - Serum Creatinine at Day 7 | Day 7
Change in Renal parameters - Serum Creatinine at Day 30 | Day 30
Change in Renal parameters - Serum Creatinine at Day 90 | Day 90
Hepatic encephalopathy: Grading as per West Haven Classification. | Day 7
  West Haven Grade (1-4) will be used to assess Hepatic Encephaloapthy, Grade 4 means worse outcome.
Hepatic encephalopathy: Grading as per West Haven Classification. | Day 30
  West Haven Grade (1-4) will be used to assess Hepatic Encephaloapthy, Grade 4 means worse outcome.
Hepatic encephalopathy: Grading as per West Haven Classification. | Day 90
  West Haven Grade (1-4) will be used to assess Hepatic Encephaloapthy, Grade 4 means worse outcome.
Proportion of participants developing Na < 120 meg/l Day 7 | Day 7
Proportion of participants developing Na < 120 meg/l Day 30 | Day 30
Proportion of participants developing Na < 120 meg/l Day 90 | Day 90
Dose of Diuretic in each arm Day 7 | Day 7
Dose of Diuretic in each arm Day 30 | Day 30
Dose of Diuretic in each arm Day 90 | Day 90
Proportion of patient developing Spontaneous Bacterial Peritonitis at Day 7 | Day 7
Proportion of patient developing Spontaneous Bacterial Peritonitis at Day 30 | Day 30
Proportion of patient developing Spontaneous Bacterial Peritonitis at Day 90 | Day 90
Proportion of patients developing Spontaneous Bacterial Empyema Day 7 | Day 7
Proportion of patients developing Spontaneous Bacterial Empyema Day 30 | Day 30
Proportion of patients developing Spontaneous Bacterial Empyema Day 90 | Day 90
No. of days pateint surviving without Liver transplant and TIPS at Day 7 | Day 7
No. of days pateint surviving without Liver transplant and TIPS at Day 30 | Day 30
No. of days pateint surviving without Liver transplant and TIPS at Day 90 | Day 90
Incidence of Post procedure complications in between both groups at Day 7 | Day 7
Incidence of Post procedure complications in between both groups at Day 30 | Day 30
Incidence of Post procedure complications in between both groups at Day 90 | Day 90
Changes in MELD between the groups | Day 7
Changes in MELD between the groups | Day 30
Changes in MELD between the groups | Day 90
Changes in CTP between the groups | Day 7
Changes in CTP between the groups | Day 30
Changes in CTP between the groups | Day 90
Number of Episodes of Hospitalization between both groups at Day 7 | Day 7
Number of Episodes of Hospitalization between both groups at Day 30 | Day 30
Number of Episodes of Hospitalization between both groups at Day 90 | Day 90
Cumulative dose of albumin at D7 in two groups | Day 7
Cumulative dose of albumin at D30 in two groups | Day 30
Cumulative dose of albumin at D90 in two groups | Day 90

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India